CLINICAL TRIAL: NCT02838589
Title: The Effect of Glucagon-like Peptide 1 (GLP-1) Receptor Agonist on Cerebral Blood Flow Velocity in Non-Stroke Volunteers (EGRABINS1)
Brief Title: The Effect of GLP-1 Receptor Agonist on Cerebral Blood Flow Velocity in Non-stroke Volunteers
Acronym: EGRABINS1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christina Kruuse (Other)
Responsible Party: Sponsor-Investigator, Christina Kruuse, MD, PhD, DMSc, Consultant Neurologist, Associate Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-16022532; 2016-001221-14 (EudraCT Number)
Record Dates: First submitted 2016-07-05; First posted 2016-07-20 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Stroke
Keywords: Cerebrovascular Stroke; Ischemic Stroke; Glucagon like peptide - 1
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Exenatide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Byetta (Active Comparator): Pre- and post treatment investigations:
  1. Mean flow velocity of the middle cerebral arteries bilateral by transcranial doppler
  2. Cerebral cortical oxygination by near infrared spectroscopy (NIRS)
  3. Endothelial function/response by the methods:
     * Biomarkers in blood (eg. e-selectin, VCAM, ICAM, endothelin, ADMA, miRNA)
     * EndoPAT2000
     * Ankle-brachial index
  Interventions: Drug: Byetta
- Isotonic saline (Placebo Comparator): Pre- and post treatment investigations:
  1. Mean flow velocity of the middle cerebral arteries bilateral by transcranial doppler
  2. Cerebral cortical oxygination by near infrared spectroscopy (NIRS)
  3. Endothelial function/response by the methods:
     * Biomarkers in blood (eg. e-selectin, VCAM, ICAM, endothelin, ADMA, miRNA)
     * EndoPAT2000
     * Ankle-brachial index
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Byetta — Single dose of subcutaneous injection of 5 μg exenatide (Byetta).
  Other Names: exenatide; GLP-1 receptor analogue; GLP-1 receptor agonist
  Arms: Byetta
Drug: Isotonic saline — Single dose of subcutaneous injection of 20 μL isotonic saline (placebo).
  Other Names: Normal saline
  Arms: Isotonic saline

SUMMARY:
This randomized controlled trial investigates the effect of a single dose of glucagon-like peptide-1 (GLP-1) receptor agonist on cerebral blood flow velocity and cortical oxygination in humans without cerebrovascular disease. This study serves as a control for a similar study investigating the effect in stroke patients (ref. to EGRABIS1).

DETAILED DESCRIPTION:
Glucagon-like peptide-1 (GLP-1) receptor agonists are widely used in the treatment of type 2 diabetes due to their ability to mimic the incretin hormone, GLP-1. GLP-1 increases glucose-dependent insulin secretion and thereby reduces plasma glucose level. Over the past few years, GLP-1 receptor agonists have been investigated as possible therapies for neurological disorders, due to their ability to cross the blood-brain-barrier. Evidence of the treatment of cerebrovascular diseases has been growing especially in animal stroke models. GLP-1 receptors, which are located in the central nervous system on neurons and endothelium, are upregulated in the brain due to ischemia. GLP-1 receptor agonists have shown anti-inflammatory and anti-apoptotic properties, and they may protect the cell from oxidative stress and may protect the endothelium. The inner lining of blood vessels, the endothelium, is an active component of the endocrine function. It affects the formation of blood clots and plays a role in the disease mechanisms of stroke. The current acute and prophylactic treatments of stroke are mainly target platelet function, but not endothelial function.

This double-blinded, randomized, controlled trial investigates the effect of a single dose of the GLP-1 receptor agonist, exenatide, on cerebral blood flow velocity, cortical oxygation and endothelial function in subjects free of cerebrovascular diseases. To our knowledge, the effect of GLP-1 receptor agonists on cerebral blood flow velocity in healthy subjects has not yet been clarified, and this study serves as a control for a similar study investigating the effect on stroke patients (ref. to EGRABIS1).

The primary endpoint is the change in mean flow velocity in the middle cerebral arteries measured by transcranial doppler. The secondary endpoints are the effects on the peripheral endothelium, hereby: 1) changes in the reactive hyperaemia index measured by EndoPAT2000, 2) changes in the ankle-brachial index, and 3) changes in endothelial/inflammatory biomarkers in the blood. The primary and secondary endpoints are measured before and up till three hours after administration of exenatide.

The overall hypothesis is that GLP-1 receptor agonists may represent a novel potential neuroprotective treatment in stroke.

ELIGIBILITY:
Inclusion Criteria:

* Person ≥ 50 years of age
* Has given written informed consent

Exclusion Criteria:

* Intracerebral haemorrhage
* Subdural / epidural hemorrhage
* subarachnoid haemorrhage
* previously major structural damage to the brain (eg. sequelae after large stroke or brain surgery)
* Diabetes type 1
* Diabetes type 2
* Known atrial fibrillation
* > 50% stenosis of internal carotid
* Known allergy to GLP-1 receptor agonists
* Hepatic impairment (ALT> 3 x upper normal limit)
* Renal impairment (eGFR <30 ml / min)
* Inflammatory bowel disease
* Previous pancreatitis
* Heart failure (NYHA class 3-4)
* Pregnancy or lactation
* Patient not expected to co-operate to the investigations
* Visualization of the middle cerebral artery bilaterally by transcranial doppler not possible

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Changes in the mean flow velocity in the middle cerebral arteries and in cortical oxigination . | Up till 3 hours
  Change in the mean flow velocity in the middle cerebral arteries will be measured with transcranial doppler and cortical oxygination by near infrared spectroscopy (NIRS) before and up till tree hours after injection of exenatide/placebo.

SECONDARY OUTCOMES:
Changes in the endothelial reactivity measured by non-invasive pletysmography. | 3 hours
  Measurement of the endothelial function by non-invasive plethysmography (EndoPAT2000) before and three hours after injection of exenatide/placebo.
Changes in the endothelial/inflammatory biomarkers in blood. | 3 hours
  Venous blood samples to measure changes in the endothelial/inflammatory biomarkers (eg. e-selectin, VCAM, ICAM, ADMA, endothelin, miRNA) before and three hours after injection of exenatide/placebo.
Changes in the ankle-brachial index. | 3 hours
  Changes in the ankle-brachial index (systolic blood pressure in ankle/arm) measured before and three hours after injection of exenatide/placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Christina R Kruuse, MD, PhD, Principal Investigator — Consultant Neurologist, Dept Neurology, Herlev Hospital
Locations (1):
- Department of Neurology, Herlev-Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olmestig J, Marlet IR, Vilsboll T, Rungby J, Rostrup E, Lambertsen KL, Kruuse C. A single dose of exenatide had no effect on blood flow velocity in the middle cerebral artery in elderly healthy volunteers: Randomized, placebo-controlled, double-blind clinical trial. Front Aging Neurosci. 2022 Jul 25;14:899389. doi: 10.3389/fnagi.2022.899389. eCollection 2022. PMID 36636739